CLINICAL TRIAL: NCT06025812
Title: A Randomized, Double-blind, Active-controlled Clinical Study Evaluating the Immunogenicity and Safety of Omicron BA.4/5-Delta Recombinant Novel Coronavirus Protein Vaccine (CHO Cells) in People Aged 18 Years and Older With Different Immunization Programs
Brief Title: Clinical Study of Omicron BA.4/5-Delta Strain Recombinant Novel Coronavirus Protein Vaccine (CHO Cells)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2023-NCV-05
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Coronavirus
Keywords: Omicron BA.4/5-Delta strain
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0-1-month immune program study group (Experimental): According to the 0-1-month immunization schedule, two doses of 25 μg/0.5 ml Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) were injected into the deltoid muscle of the upper arm.
  Interventions: Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells)
- 0-1-month immune program control group (Active Comparator): According to the 0-1-month immunization schedule, two doses of 25 μg/0.5 ml recombinant novel coronavirus protein vaccine (CHO cells) were injected into the deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant novel coronavirus protein vaccine (CHO cells)
- 0-6-month immune program study group (Experimental): The subjects were from the "LKM-2023-NCV-02" project and were vaccinated on a voluntary basis with 25 μg/0.5 ml Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) at the visit 6 months after the exemption.
  Interventions: Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells)
- 0-6-month immune program control group (Active Comparator): The subjects were from the "LKM-2023-NCV-02" project and were vaccinated on a voluntary basis with 25 μg/0.5 ml recombinant novel coronavirus protein vaccine (CHO cells) at the visit 6 months after the exemption.
  Interventions: Biological: Recombinant novel coronavirus protein vaccine (CHO cells)

INTERVENTIONS:
Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells).
  Arms: 0-1-month immune program study group; 0-6-month immune program study group
Biological: Recombinant novel coronavirus protein vaccine (CHO cells) — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose Recombinant new coronavirus vaccine (CHO cells).
  Arms: 0-1-month immune program control group; 0-6-month immune program control group

SUMMARY:
Popular title: Clinical study of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells).

Purpose of the study: Main objectives: To evaluate the immunogenicity and safety of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) against the new coronavirus prototype strain and Omicron variant (XBB, BA.5, BF.7) after receiving 2 doses according to different immunization schedules in people aged 18 years and older. Secondary purposes: To evaluate the immune persistence of Omicron BA.4/5-Delta recombinant novel coronavirus protein vaccine (CHO cells) against the new coronavirus prototype strain and Omicron variant (XBB, BA.5, BF.7) after receiving 2 doses according to different immunization schedules in people aged 18 years and older.

Overall design: Studies were randomized, double-blind, active-controlled study design.

Study group: There were 160 participants aged 18 years and older, including 80 people aged 60 years and older.

Study group：Among them, 80 subjects were from the "randomized, double-blind, active-controlled clinical study to evaluate the immunogenicity and safety of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) in people aged 18 years and older, protocol number: LKM-2023-NCV-02", 40 cases in the study group and 40 cases in the control group, and completed the second dose of vaccine at the 6th month visit to observe immunogenicity and safety. The remaining 80 subjects were randomly blinded to the 1:1 ratio into the research group and the control group and received 2 doses of the experimental vaccine according to the 0-1-month procedure to observe immunogenicity and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older at the time of signing the informed consent form.
2. The subject himself voluntarily participates in the study, signs the informed consent form, and can provide legal identification, understand and comply with the requirements of the research protocol.
3. More than 6 months after completing the basic immunization or booster immunization of the new coronavirus vaccine.
4. Female subjects of childbearing age and male subjects who were able to use effective contraception during the study.

Exclusion Criteria:

Participants were not eligible for study if they had any of the following:

1. Previous history of severe allergy to any vaccine, or history of severe allergy to any component of the study vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, Henoch-Schönlein purpura, thrombocytopenic purpura, dyspnea, angioedema, allergic constitution (such as allergy to two or more drugs, food or pollen), etc.
2. fever (axillary body temperature≥ 37.3°C) within 72 hours before enrollment, or axillary body temperature ≥ 37.3°C on the day of enrollment.
3. Patients infected with the new coronavirus within 3 months before enrollment (asymptomatic infection or positive nucleic acid or antigen test of the new coronavirus).
4. Patients with aplastic anemia that has not been relieved, primary immune thrombocytopenia (ITP) active period, and uncontrolled coagulation diseases.
5. history of congenital or acquired immunodeficiency or autoimmune disease; no history of spleen or spleen surgery or trauma; or receive immunomodulators within 6 months, such as corticosteroids in immunosuppressant doses (dose reference: equivalent to prednisone 20 mg/day for more than one week); or monoclonal antibodies; or thymus peptide; or interferon, etc.; However, topical medications (such as ointments, eye drops, inhalers, or nasal sprays) are allowed; Lymphoproliferative disorders are not controlled.
6. Non-live vaccine ≤ 14 days before vaccination and live attenuated vaccine 30 days before ≤vaccination.
7. Patients with malignant tumors who are undergoing chemotherapy, radiotherapy, immunotherapy, etc. before and after surgery, Patients in the state of organ transplantation.
8. Those suffering from uncontrolled epilepsy and other progressive neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.).
9. Patients with acute diseases, or acute exacerbations of chronic diseases, or uncontrolled severe chronic diseases, such as hypertension that cannot be controlled by drugs (systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥100mmHg).
10. Lactating women or pregnant women; The investigator believes that the participant has any disease or condition that would put the participant at risk, the participant cannot complete the study as required by the protocol, and there are circumstances that interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events after 2 doses given intramuscularly according to different immunization programs | 6 months after 2 doses of vaccine
  The observation of adverse events mainly come from vital sign detection and laboratory examination (including blood routine/urine routine/blood biochemistry/electrocardiogram and chest X-ray), local reactions and systemic reactions after injection.
Laboratory markers of immunity after 2 doses given intramuscularly according to different immunization programs | 14 days after 2 doses of vaccine
  Geometric mean titer (GMT) of neutralizing antibodies against the Omicron variant (XBB) after vaccination with the investigational vaccine.
Immunogenic end points | 14 days after 2 doses of vaccine
  Positive conversion rate of the Omicron variant (XBB) of the new coronavirus after vaccination with the investigational vaccine.

SECONDARY OUTCOMES:
Laboratory markers of immunity | 14 days after 2 doses of vaccine
  Geometric mean titer (GMT) of neutralizing antibodies against the prototype novel coronavirus strain, Omicron strain (BA.4/5, BF.7) after 2 doses of vaccine candidate.
Laboratory markers of immunity | 14 days after 2 doses of vaccine
  Growth multiples (GMI) of the prototype new coronavirus strain and the Omicron variant (BA.4/5, BF.7) after 2 doses of investigational vaccine.
Immunogenic end points | 14 days after 2 doses of vaccine
  Positive conversion rate against the prototype Omicron variant (BA.4/5, BF.7) after 2 doses of study vaccine.
Laboratory markers of immunity | 14 days after 2 doses of vaccine
  Growth multiple (GMI) of the new coronavirus Omicron variant (XBB) after 2 doses of investigational vaccine.
Laboratory markers of immunity | 6 months after 2 doses of vaccine
  Geometric mean titer (GMT) of neutralizing antibodies against the prototype novel coronavirus strain, Omicron strain (XBB, BA.4/5, BF.7) after 2 doses of vaccine candidate.
Laboratory markers of immunity | 6 months after 2 doses of vaccine
  Growth multiples (GMI) of the prototype new coronavirus strain and the Omicron variant (XBB, BA.4/5, BF.7) after 2 doses of investigational vaccine.
Immunogenic end points | 6 months after 2 doses of vaccine
  Positive conversion rate against the prototype Omicron variant (XBB, BA.4/5, BF.7) after 2 doses of study vaccine.